CLINICAL TRIAL: NCT04283422
Title: Diagnosis of Lower Respiratory Tract Infections in Pediatric Patients in Intensive Care Unit Using Biofire Filmarray
Brief Title: Diagnosis of Lower Respiratory Tract Infections Using Biofire Filmarray
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Kadry Moawad, assistant lecturer, Assiut University
Other Study IDs: Biofire filmarray in LRTI
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Biofire Filmarray

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patintes on mechanical ventilation
  Interventions: Diagnostic Test: Biofire filmarray
- patintes not on mechanical ventilation
  Interventions: Diagnostic Test: Biofire filmarray

INTERVENTIONS:
Diagnostic Test: Biofire filmarray — Identification of microorganisms including:
  1. Isolation of microorganisms:
     The sample will be cultured on blood agar, chocolate agar , MacConkeys agar and Sabouraud dextrose agar (SDA) plates,
  2. Identification of the organism by Vitek2
  3. Antibiotic sensitivity test of the organism by Vitek2
  4. Identification of the organism by Biofire filmarray
  Other Names: Vitek2

SUMMARY:
Comparison of pathogens causing lower respiratory tract infections in ventilated versus non ventilated pediatric patients in intensive care unit using biofire filmarray and vitek2

* Antibiotic sensitivity using vitek2
* Comparison of the type of antibiotic resistance using biofire filmarray and vitek2
* To provide information about prevalence of these organisms.

DETAILED DESCRIPTION:
Acute respiratory infections (ARI) are a leading cause of morbidity and mortality worldwide. Although usually more severe in children, the elderly and immunocompromised patients, all populations and age groups are susceptible.

Lower respiratory infections are the third leading cause of death worldwide and nearly two million childhood deaths worldwide are attributable to ARI, with the vast majority occurring in developing countries.The World Health Organization estimates that in 2013, over 8% of all deaths in the Eastern Mediterranean Region were attributable to ARIs. However, regional data on morbidity and etiology of these infections are lacking.

These infections have a significant impact on antimicrobial prescriptions, hospitalizations and lost time from work and school. The most frequent agents responsible for ARI are respiratory viruses followed by bacteria .Empiric treatment with antibiotics is frequently initiated even when viral infection is a strong possibility,leading to unnecessary antibiotic use . The early diagnosis of the pathogen is beneficial for the precise selection of medication,which can largely avoid the overuse or even abuse of the antibiotics and improve the clinical care of patients. More importantly, the early diagnosis of contagious pathogens, such as Bordetella pertussis (B. pertussis) and influenza viruses, can enable early isolation of patients, thus reducing the spread of pathogens.

At present, the routine detection methods for respiratory pathogens are mostly based on immunological methods.

Direct diagnosis of respiratory viruses by antigen detection using immunofluorescence assays (IFA), is still used but is typically limited to eight viruses (adenovirus [AdV], influenza A [FluA], influenza B [FluB], parainfluenza [PIV], human metapneumovirus [HMPV] and respiratory syncytial virus [RSV]) and may lack sensitivity depending on the viral titer, patient´s age and time of testing in relation to the onset of symptoms .

Molecular methods such as Polymerase chain reaction (PCR) increase viral detection due to a greater analytic sensitivity compared to conventional methods such as antigen detection and/or viral culture.

Microbiological analysis and identification of organisms may take 48-72 h,false negative results may occur as a result of concomitant or previous antibiotic treatment , whereas false positive may represent colonization or sampling errors.

The VITEK 2 is a fully automated system for microbial identification and antimicrobial susceptibility testing (AST ), after a primary inoculums has been prepared and standardized . With its colorimetric reagent cards, the VITEK 2 offers a state of the art technology platform for phenotypic identification methods.(6) The application of FilmArray respiratory panel in the diagnosis of lower respiratory tract infections is designed to reduce the time for identification of the microorganisms FilmArray is a small, desktop, fully automated multiplex PCR device. The molecular system includes automated nucleic acid extraction, an initial reverse transcription step and multiplex nested PCR, followed by a melting curve analysis .

The BIOFIRE® FILMARRAY® Pneumonia Panel plus tests for 18 bacteria (11 Gram negative, 4 Gram positive and 3 atypical), 7 antibiotic resistance markers, and 9 viruses that cause pneumonia and other lower respiratory tract infections. It offers an overall sensitivity and specificity for bronchoalveolar (BAL)-like samples of 96,2% and 98.3%, respectively, and for sputum samples a sensitivity and specificity of 96.3% and 97.2%, respectively.The test is performed in a closed system that requires 5 min of hands-on time and 65 min of instrumentation time. Several comparison studies between FilmArray and other tests for respiratory organisms showed comparable results .

ELIGIBILITY:
Inclusion Criteria:

- Pediatric patients with acute lower respiratory tract infections.

Exclusion Criteria:

* Age above 18 years old

Ages: 10 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with acute lower respiratory tract infections.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of pathogens causing lower respiratory tract infections in ventilated versus non ventilated pediatric patients in intensive care unit | one year
  Percentage of pathogens including viruses ,bacteria and fungi responsible for lower respiratory tract infections will be carried out by using biofire Filmarray and vitek 2
Prevalence of drug resistance in bacteria | one year
  Gene of drug resistance in bacteria will be detected by using biofire Filmarray and phenotypic tests by using vitk2 vitek2
prevalence of pathogens causing lower respiratory tract infections . | one year
  prevalence of both bacterial and fungal infection causing lower respiratory tract infections by vitek2

SECONDARY OUTCOMES:
Rapid identification of causative organisms in critical cases. | one hour
  Rapid identification of causative organisms in critical cases bu using the biofire filmarray

REFERENCES:
- [Background] Rowlinson E, Dueger E, Mansour A, Azzazy N, Mansour H, Peters L, Rosenstock S, Hamid S, Said MM, Geneidy M, Abd Allah M, Kandeel A. Incidence and etiology of hospitalized acute respiratory infections in the Egyptian Delta. Influenza Other Respir Viruses. 2017 Jan;11(1):23-32. doi: 10.1111/irv.12409. Epub 2016 Aug 12. PMID 27458989
- [Background] Li J, Tao Y, Tang M, Du B, Xia Y, Mo X, Cao Q. Rapid detection of respiratory organisms with the FilmArray respiratory panel in a large children's hospital in China. BMC Infect Dis. 2018 Oct 11;18(1):510. doi: 10.1186/s12879-018-3429-6. PMID 30305033
- [Background] Chun K, Syndergaard C, Damas C, Trubey R, Mukindaraj A, Qian S, Jin X, Breslow S, Niemz A. Sepsis Pathogen Identification. J Lab Autom. 2015 Oct;20(5):539-61. doi: 10.1177/2211068214567345. Epub 2015 Jan 28. PMID 25631157
- [Background] Wahrenbrock MG, Matushek S, Boonlayangoor S, Tesic V, Beavis KG, Charnot-Katsikas A. Comparison of Cepheid Xpert Flu/RSV XC and BioFire FilmArray for Detection of Influenza A, Influenza B, and Respiratory Syncytial Virus. J Clin Microbiol. 2016 Jul;54(7):1902-1903. doi: 10.1128/JCM.00084-16. Epub 2016 Apr 20. PMID 27098956